CLINICAL TRIAL: NCT05148988
Title: Feasibility of Ultrasound Particle Image Velocimetry to Quantify Flow in the Abdominal Aorta Before and After Endovascular Aneurysm Repair
Brief Title: Ultrasound Velocimetry in the Abdominal Aorta Before and After Endovascular Aneurysm Repair
Acronym: EchoPIV in AAA
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: University of Twente (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1917
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AAA patients: The entire cohort consists of patients with an abdominal aortic aneurysm eligible for endovascular repair using an Endurant II device.
  Interventions: Diagnostic Test: EchoPIV; Diagnostic Test: 4D flow MRI

INTERVENTIONS:
Diagnostic Test: EchoPIV — All patients will undergo an echoPIV measurement 6 to 8 weeks before and 6 to 8 weeks after endovascular aneurysm repair. These measurements will take place at the Vascular Center of Rijnstate Hospital. A venous cannula will be inserted to enable contrast administration. Ultrasound data will be collected at the caudal renal artery, infrarenal neck, aneurysm sac and both iliac arteries.
Diagnostic Test: 4D flow MRI — A 4D phase-contrast magnetic resonance imaging (4D flow MRI) scan of the abdominal aorta will be obtained 6 to 8 weeks before and 6 to 8 weeks after endovascular aneurysm repair.

SUMMARY:
Rationale: An abdominal aortic aneurysm (AAA) is a common vascular disease with a high mortality in case of rupture. The underlying processes initiating aneurysmal degeneration and driving aneurysmal growth remain poorly understood. Local hemodynamics might play a key role in the pathogenesis of AAA, as it is associated with aneurysmal growth, intraluminal thrombus formation and rupture risk. Visualizing and quantifying local blood flow profiles could eventually provide more insight in the underlying mechanisms of aneurysm progression as well as identify smaller AAA with increased vulnerability or larger AAA with low risk of rupture. Consequently, this may improve risk assessment and provide patient-specific therapy guidance. Nowadays, endovascular aneurysm repair (EVAR) is the preferred treatment modality in most patients with an infrarenal AAA. However, EVAR is associated with a relatively high reintervention rate. It is hypothesized that the placement of a stent graft may alter local hemodynamics and subsequent recirculations or flow stagnations promote the onset of thrombosis or micro-emboli. These unfavourable flow conditions might be related to various complications after EVAR, such as limb occlusion, renal dysfunction, and the persistence of type II endoleaks. Visualizing local blood flow profiles after EVAR might provide insight in these (un)favourable conditions. In vivo blood flow quantification is a great challenge, particularly in the abdomen. Advanced ultrasound based techniques, incorporating ultrasound contrast agents and plane wave imaging, proved to be feasible in quantifying aortoiliac blood flow patterns in healthy volunteers.

Objective: The aim of this study is to determine the feasibility of ultrafast contrast-enhanced ultrasound particle image velocimetry (echoPIV) measurements to quantify spatiotemporal blood flow velocity profiles in the abdominal aorta of AAA patients before and after endovascular repair.

Secondary objectives are to determine the correlation between echoPIV and phase-contrast MRI (PC MRI) based measurements to ultimately validate the spatiotemporal velocity profiles obtained with echoPIV. Furthermore, changes in blood flow velocity profiles after placement of a stent graft will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age
* BMI ≤ 30 kg/m2
* Infrarenal AAA
* Scheduled for elective EVAR with the Endurant II stent graft
* Informed consent form understood and signed, and agrees to all visits

Exclusion Criteria:

* Hypersensitivity to the active substance(s) or any of the excipients in Sonovue
* Right-to-left cardiac shunt
* Severe pulmonary hypertension (pulmonary artery pressure > 90mmHg)
* Uncontrolled systemic hypertension
* Severe pulmonary disease (e.g. COPD GOLD 3 or 4, adult respiratory distress syndrome)
* Clinically unstable cardiac disease (recent, < 3 months, or ongoing myocardial infarction, unstable angina at rest, recent percutaneous coronary intervention, clinically worsening cardiac symptoms, severe cardiac arrhythmia's, endocarditis, etc.)
* Prosthetic valves
* Loss of renal function (GFR < 31 ml/min), end-stage renal disease
* End-stage liver disease
* Sepsis
* Hypercoagulable status, recent (< 3 months) thrombosis
* Congestive heart failure (class III or IV)
* Pregnancy
* MRI exclusion criteria (pacemakers, cerebral vascular clips, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an abdominal aortic aneurysm eligible for endovascular repair using the Endurant II device.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment vector velocity fields | 6 to 8 weeks after the procedure (endovascular repair)
  Vector velocity fields derived from the echoPIV data will be used to calculate and visualize the velocity profile. In order to answer the question regarding feasibility of echoPIV the quality of the vector velocity fields will be assessed using three different metrics of which the first one is a qualitative assessment by different observers. Recordings of the contrast-enhanced ultrasound with an overlay of the vector velocity profiles will be reviewed on different topics following a scoring rubrics.
Contrast-to-background ratio | 6 to 8 weeks after the procedure (endovascular repair)
  The contrast-to-background ratio (CBR) is the second metric to assess the outcomes of the echoPIV measurements. The CBR is a quantitative measure for the contrast levels and therefore for the quality of the contrast-enhanced US image. The higher the CBR level (in dB) the higher the intensity of the contrast which is needed for sufficient PIV analysis.
Vector correlation | 6 to 8 weeks after the procedure (endovascular repair)
  The vector correlation is the third metric to assess the outcomes of the echoPIV measurements. The vector correlation demonstrates the tracking performance of the PIV algorithm. The vector correlation provides a unitless value between 0 and 1 in which 0 indicates poor tracking of the microbubble contrast and 1 indicates perfect tracking of the microbubble contrast.

SECONDARY OUTCOMES:
Correlation echoPIV and 4D flow MRI | 6 to 8 weeks after the procedure (endovascular repair)
  EchoPIV derived local hemodynamics will be compared to outcomes of the 4D flow MRI scan.
Influence of stent-graft placement | 6 to 8 weeks after the procedure (endovascular repair)
  EchoPIV derived local hemodynamics prior to- and after placement of the stent-graft will be compared.
Vorticity | 6 to 8 weeks after the procedure (endovascular repair)
  Multiple blood flow parameters will be derived from the echoPIV data. The first one is the vorticity, or the curl of the velocity. The vorticity represents the rotation of particles inside the flow field. This measure can potentially be used to define regions with disturbed blood flow, as a high value (in rad/s) indicates the occurence of a recirculation.
Vector complexity | 6 to 8 weeks after the procedure (endovascular repair)
  The second blood flow parameters derived from the echoPIV data is the vector complexity. Vector complexity is a measure of multi-directional flow, ranging from 0 till 1. a value of 1 means complex flow with all velocity vectors pointing in all directions, whereas a value of 0 means laminar flow with all velocity vectors pointing in the same direction. This measure can potentially be used to indicate regions with disturbed blood flow.

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands